CLINICAL TRIAL: NCT04589754
Title: An Open, Multi-center, Randomized, Phase II Study of Adriamycin and Ifosfamide Combined With Sintilimab in the Treatment of Advanced or Unresectable Soft Tissue Sarcoma
Brief Title: Adriamycin and Ifosfamide Combined With Sintilimab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xing Zhang, Director of department of medical sarcoma and melanoma,Principal Investigator,Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sintilimab plus chemotherapy
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — sintilimab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab plus chemotherapy (Experimental): Adriamycin and ifosfamide combined with sintilimab in the treatment of advanced or unresectable soft tissue sarcoma
  Interventions: Drug: Sintilimab plus chemotherapy; Drug: Adriamycin-based chemotherapy
- Adriamycin-based chemotherapy (Placebo Comparator): Adriamycin-based chemotherapy in the treatment of advanced or unresectable soft tissue sarcoma
  Interventions: Drug: Sintilimab plus chemotherapy; Drug: Adriamycin-based chemotherapy

INTERVENTIONS:
Drug: Sintilimab plus chemotherapy — AI regimen chemotherapy (ADM 50 mg / m2, D1 + IFO 2.5 g / m2, D1-3, IV drip) was used for 3 weeks; CAV / IE regimen alternate chemotherapy (regimen 1: CTX 1.2mg/m2 D1 + ADM 50mg / m2 D1 + VCR 1.4mg/m2 D1 and regimen 2: IFO 1.5g/m2 D1-5 + VP-16 100mg / m2 D1-5, IV drip). Regimen 1 and 2 were performed alternately, with a cycle of 3 weeks; sintilimab (10ml; 100mg) was administered intravenously every 3 weeks.
Drug: Adriamycin-based chemotherapy — AI regimen chemotherapy (ADM 50 mg / m2, D1 + IFO 2.5 g / m2, D1-3, IV drip) was used for 3 weeks; CAV / IE regimen alternate chemotherapy (regimen 1: CTX 1.2mg/m2 D1 + ADM 50mg / m2 D1 + VCR 1.4mg/m2 D1 and regimen 2: IFO 1.5g/m2 D1-5 + VP-16 100mg / m2 D1-5, IV drip). Regimen 1 and 2 were performed alternately, with a cycle of 3 weeks.

SUMMARY:
The aim of this study was to explore the efficacy and safety of adriamycin and ifosfamide combined with sintilimab versus chemotherapy in the treatment of advanced or unresectable soft tissue sarcoma.

DETAILED DESCRIPTION:
At present, there are a number of clinical trials of chemotherapy drugs combined with anti PD-1 antibody in the treatment of cancer, but the clinical research of chemotherapy containing adriamycin combined with anti-PD-1 antibody for advanced STS patients is almost blank. Regimen containing adriamycin is the standard chemotherapy regimen for advanced STS approved by international guidelines. As an innovative PD-1 monoclonal antibody, more phase II clinical studies are needed to evaluate the efficacy and safety of sintilimab in a variety of cancers. For patients who fail or cannot tolerate first-line treatment, treatment options are still limited. In view of the above problems, this study aims to observe and explore the efficacy and safety of chemotherapy including adriamycin combined with sintilimab versus chemotherapy in the second-line treatment of patients with advanced STS, so as to provide more and better treatment options for patients with advanced STS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in the study and signed informed consent;

   All advanced or non resectable soft tissue sarcomas confirmed by pathology failed or did not have standard treatment or could not tolerate standard treatment, Have at least one according to RECIST 1.1 the standard measurable lesions mainly included synovial sarcoma, leiomyosarcoma, alveolar soft tissue sarcoma, undifferentiated pleomorphic sarcoma / malignant fibrous histiocytoma, liposarcoma, fibrosarcoma, clear cell sarcoma, angiosarcoma, epithelioid sarcoma, malignant peripheral nerve sheath tumor, undifferentiated sarcoma, dermatofibrosarcoma protuberans, inflammatory myofibroblastic sarcoma Malignant solitary fibroma, sarcoma after radiotherapy. However, there are no standard treatment types, such as alveolar soft tissue sarcoma, post radiotherapy sarcoma, highly differentiated / dedifferentiated / pleomorphic liposarcoma, clear cell sarcoma, etc.; except for the following types: chondrosarcoma, osteosarcoma, malignant mesothelioma, gastrointestinal stromal tumor, etc;
2. Advanced patients with unresectable lesions or lymph nodes or distant metastasis assessed by imaging;
3. In the past three months, there was at least one measurable target lesion according to RECIST version 1.1 standard, and it can be accurately measured by magnetic resonance imaging (MRI) or computer tomography (CT) in at least one direction (the maximum diameter needs to be recorded), with conventional CT ≥ 20 mm or spiral CT ≥ 10 mm.
4. They were 14-70 years old; ECoG PS score: 0-1; the expected survival time was more than 3 months;
5. Within 7 days before treatment, the main organ functions met the following criteria:

(1) Blood routine examination standard (without blood transfusion within 14 days)

① Hemoglobin (HB) ≥ 90g / L;

② The absolute value of neutrophil (ANC) ≥ 1.5 × 109 / L;

* Platelet (PLT) ≥ 80 × 109 / L.

  (2) Biochemical examination should meet the following standards:

  ① Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN);

  ② Alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5uln, such as

With liver metastasis, ALT and AST ≤ 5uln;

③ Serum creatinine (CR) ≤ 1.5uln or creatinine clearance rate (CCR) ≥ 60ml / min;

(3) Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ the lower limit of normal value (50%).

Women of childbearing age should agree that contraceptive measures (such as intrauterine device, contraceptive or condom) must be used during the study period and within 6 months after the end of the study; serum or urine pregnancy test negative within 7 days before study enrollment, and must be non lactating patients; men should agree that contraceptive measures must be used during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

1) Patients who had previously received anti-PD-1 / PD-L1 antibody therapy.

2) Other malignancies occurred or were present within 5 years, except for cervical carcinoma in situ, non melanoma skin cancer and superficial bladder tumor [ta (non invasive tumor), tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];

3) The patients with thyroid dysfunction after the best drug treatment;

4) Systemic anti-tumor therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or mitomycin C within 6 weeks prior to the trial drug treatment) was planned within 4 weeks before enrollment or during the study period. Over extended field radiotherapy (ef-rt) was performed within 4 weeks before admission or limited field radiotherapy (rfrt) was performed within 2 weeks before grouping;

5) With pleural effusion or ascites, it causes respiratory syndrome (≥ CTC AE grade 2 dyspnea [grade 2 dyspnea refers to shortness of breath with a small amount of activity; it affects instrumental activities of daily living]);

6) Any unrelieved toxic reaction higher than CTC AE (4.01) grade 1 or above caused by previous treatment, excluding alopecia;

7) Patients with any severe and / or uncontrolled disease, including:

1. Patients with poor blood pressure control (SBP ≥ 150 mmHg, DBP ≥ 100 mmHg);
2. Patients with myocardial ischemia or myocardial infarction of grade I or above, arrhythmia (including QTc ≥ 480ms) and congestive heart failure (NYHA) grade ≥ 2;
3. Active or uncontrolled severe infection (≥ CTC AE Level 2 infection);
4. Chronic liver disease, decompensated liver disease or decompensated hepatitis;
5. Renal failure needs hemodialysis or peritoneal dialysis;
6. Poor control of diabetes mellitus (FBG > 10mmol / L);
7. Urine routine examination showed that urine protein was ≥ + +, and 24-hour urine protein was more than 1.0 G;
8. Patients with epilepsy and need treatment;

8) Major surgical treatment, open biopsy or obvious traumatic injury were performed within 28 days before admission;

9) Patients with any physical signs or history of bleeding regardless of severity; patients with any bleeding or bleeding events ≥ CTCAE 3 within 4 weeks before enrollment had unhealed wounds, ulcers or fractures;

10) Patients who had AVT events within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism;

11) There were active ulcer, intestinal perforation and intestinal obstruction;

12) Subjects with clinical symptoms of central nervous system metastasis (such as brain edema, need for hormone intervention, or brain metastasis progression); patients who have previously received treatment for brain or meningeal metastasis, such as clinical stability (MRI) for at least 2 months, and who have stopped systemic hormone therapy (dose > 10mg / day, prednisone or other effective hormones) for more than 2 weeks can be included;

13) The subjects were using immunosuppressive agents, or systemic or absorbable local hormone therapy to achieve the purpose of immunosuppression (dosage > 10mg / D, prednisone or other effective hormones), and continued to use them within 2 weeks before enrollment;

14) Subjects with any active autoimmune disease or history of autoimmune diseases (e.g., but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; if the subject has vitiligo or asthma has been completely relieved in childhood, it is not necessary to be an adult Any intervention can be included; asthma patients who need bronchodilator for medical intervention cannot be included);

15) The subjects had active tuberculosis;

16) According to the judgment of the researcher, the subjects are not suitable to be enrolled or there are other factors that may lead to termination of the study, such as other serious diseases (including mental diseases) requiring combined treatment, serious laboratory examination abnormalities, and family or social factors, which will affect the safety of the subjects, or the collection of test data and samples;

17) Patients who participated in other clinical trials of anti-tumor drugs within 28 days before enrollment.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate, ORR | up to 24 months
  The percentage of patients with complete remission and partial remission in patients with evaluable curative effect.

SECONDARY OUTCOMES:
Progression-free survival, PFS | From the beginning of observation to the end of observation（1 year) of the last enrolled patient
  PFS was defined as the time from randomization to objective tumor progression or death.
Disease-free surviva, DFS | From the beginning of observation to the end of observation (1 year) of the last enrolled patient
  DFS is defined as the time from randomization to recurrence of tumor or death.
Overall survival, OS | From the beginning of observation to the end of observation (1 year) of the last enrolled patient
  OS is defined as the time from randomization to death.

CONTACTS AND LOCATIONS:
Overall Officials: Xing Zhang, Principal Investigator — Sun Yat-sen University CancerCenter
Locations (1):
- Xing Zhang, Guangzhou, Guangdong, China